CLINICAL TRIAL: NCT06094543
Title: Improving Overactive Bladder Treatment Access and Adherence Through Personalized Behavioral Modifications and Mobile Technology-Based Interventions
Brief Title: Improving Overactive Bladder Treatment Access and Adherence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ekene Enemchukwu, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 72487
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Overactive Bladder Syndrome; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Engagement Tool (PET) (Experimental): Participants will use the PET weekly for 12 weeks
  Interventions: Behavioral: Patient Engagement Tool
- Usual Care (No Intervention): Usual Clinic Follow up every 6 weeks for 12 weeks

INTERVENTIONS:
Behavioral: Patient Engagement Tool — 8 week daily patient education and engagement tool
  Arms: Patient Engagement Tool (PET)

SUMMARY:
Overactive bladder (OAB) and urinary incontinence (UI) are chronic debilitating and embarrassing conditions that affect 33 million Americans. Yet, both are underdiagnosed and undertreated with significant financial and health-related consequences. OAB syndrome is characterized by urinary urgency, with and without urinary incontinence, urinary frequency, and nocturia. Evidence-based treatments are available, including behavioral therapy, pharmacotherapy, and minimally invasive procedures. Diagnosis and treatment are also associated with improvement in urinary symptoms and overall quality of life (QOL).3 However, 70-80% of treated patients will discontinue use of therapy in the first year due to one of several factors (e.g., cost, tolerability, inadequate effect). In addition, only 4.7% progress to advanced therapies suggesting undertreatment for those that need it most. Vulnerable populations are especially at risk, as therapy utilization are lowest among older, lower income, and/or minority groups. Poor access, insufficient patient education regarding disease chronicity, expected outcomes, costs, and potential side effects lead to unrealistic patient perceptions about therapy. This leads to suboptimal therapy duration, poor treatment efficacy, adherence, and undertreatment. The study aims to evaluate a tailored patient-centered tool to begin the treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 years or older
* OAB symptoms for at least 3 months
* English/Spanish language skills and cognitive status sufficient to complete all study related materials
* Behavioral treatment naïve patients
* Previously treated OAB patients without supervised pelvic floor physical therapy or pharmacotherapy within 1 year

Exclusion Criteria:

* Post void residual urine > 150ml
* Confirmed diagnosis of Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS)
* Pregnant or breastfeeding patients
* Patients residing in a nursing home
* Comorbid neurological conditions, including spinal cord injury, progressive neurologic illnesses (e.g. Multiple Sclerosis, Parkinson's disease) or central nervous system disease (e.g. brain tumor, stroke)
* Stage 2 or greater pelvic organ prolapse
* Any history of urethral stricture
* Any history of pelvic irradiation
* Any history of bladder malignancy
* Current symptomatic urinary tract infection (UTI), unresolved by the time of enrollment
* Hematuria without a clinical evaluation
* History or current use of indwelling urinary foley catheterization, suprapubic tube or intermittent catheterization
* Patients with UI treated with onabotulinumtoxinA, sacral neuromodulation, or percutaneous tibial nerve stimulation (third line therapies)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Systems Usability Scale (SUS) | 12 weeks
  Usability, engagement, Patient engagement tool reliability/accessibility (technical issues)
Bladder Health Knowledge, Attitudes, and Beliefs (KAB) | 12 weeks
  Will assess knowledge about bladder health
  1. Knowledge: Awareness and understanding of normal bladder function, signs and symptoms of dysfunction (e.g., incontinence, urgency), and available treatment or prevention strategies.
  2. Attitudes: Perceptions and feelings toward bladder health, such as embarrassment, stigma, or normalization of symptoms like leakage or urgency.
  3. Beliefs: Individual or cultural beliefs about the causes, severity, and treatability of bladder problems, which may influence care-seeking behavior.

SECONDARY OUTCOMES:
Therapy adherence | 12 weeks
Global Perceptions and Satisfaction with Treatment (LURN) | 12 weeks
  OAB management satisfaction
ICIQ-UI & ICIQ-OAB Combined Questionnaire | 12 weeks
  Will be used to assess change in symptom severity from baseline, 4 weeks and at 12 weeks
Self-Efficacy for Managing Chronic Conditions Questionnaire (PROMIS) | 12 weeks
  A validated patient-reported outcome measure developed by the NIH PROMIS initiative.
  The Self-Efficacy for Managing Chronic Conditions - Managing Symptoms subdomain was modified to assess a patient's confidence in their ability to monitor and manage bothersome symptoms related to chronic urinary incontinence and overactive bladder (OAB). It evaluates perceived ability to recognize symptom triggers, implement behavioral or lifestyle adjustments, and manage urinary urgency, frequency, or leakage in daily life.
  Higher scores indicate stronger self-efficacy, which has been associated with better adherence to treatment strategies, such as bladder training, fluid management, and pelvic floor exercises, in patients with OAB and incontinence.
  Each item is scored on a 5-point Likert scale with higher scores indicating greater self-efficacy. It is widely used in both clinical and research settings to assess readiness for self-management and tailor interventions accordingly.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Pelvic Health Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No